CLINICAL TRIAL: NCT06889532
Title: SAVE Studie- SArcoma Surgery With Vacuum Enhanced Wound Treatment Randomised Controlled Study to Evaluate the Wound Management in Sarcoma Surgery
Brief Title: SAVE Studie- SArcoma Surgery With Vacuum Enhanced Wound Treatment Randomised Study to Evaluate the Wound Management in Sarcoma Surgery
Acronym: SAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Maastricht University Medical Center (Other); University Hospital, Basel, Switzerland (Other); University Hospital Erlangen (Other); Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-101270-BO-ff
Record Dates: First submitted 2025-02-23; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Soft Tissue Sarcoma (STS)
Keywords: randomized; controlled; vacuum therapy; sarcoma; soft tissue sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: The study, "SAVE Study - SArcoma Surgery with Vacuum Enhanced Wound Treatment," is a prospective, ran-domized, controlled clinical trial aimed at comparing the effectiveness of two surgical approaches to optimize wound care following sarcoma resections. The study is designed as a multicenter trial.
  The study includes two arms:
  * Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days.
  * Control Group: In this group, wound closure is performed using primary sutures or staples, combined with the placement of a subcutaneous Redon drainage system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days.
  Interventions: Procedure: Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days.
- Control Group (No Intervention): Control Group: In this group, wound closure is performed using primary sutures or staples, combined with the placement of a subcutaneous Redon drainage system.

INTERVENTIONS:
Procedure: Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days. — Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to evaluate local complications following sarcoma resection in the groin and thigh regions with regard to the planned wound closure method. To this end, temporary soft tissue coverage using a vacuum-assisted closure (VAC) system and delayed secondary closure with wound sutures and drainage placement will be compared to primary closure with drainage in terms of wound infections, revisions, and seroma formation.

DETAILED DESCRIPTION:
The study, "SAVE Study - SArcoma Surgery with Vacuum Enhanced Wound Treatment," is a prospective, ran-domized, controlled clinical trial aimed at comparing the effectiveness of two surgical approaches to optimize wound care following sarcoma resections. The study is designed as a multicenter trial.

The study includes two arms:

* Intervention Group: In this group, a vacuum-assisted closure (VAC) system is applied intraoperatively to seal the wound, followed by a secondary closure after 3-7 days.
* Control Group: In this group, wound closure is performed using primary sutures or staples, combined with the placement of a subcutaneous Redon drainage system.

The planned study start date is November 1, 2024. Before enrolling patients, all participating centers must have received approval from their ethics committees.

Initially, potential participants will be assessed for eligibility based on the inclusion and exclusion criteria. They will be educated about the study and provided with a standardized information sheet across all centers. After consent, they will be enrolled in the study.

Next, patients will be randomly assigned to one of the study groups (Intervention group or Control group). This will be done through computer-assisted randomization to ensure the assignment is both random and balanced. The randomization process will be completed intraoperative after assessing the wound cavity (both wound clo-sures should be feasible).

The surgical care should be performed by a certified sarcoma surgeon. The guidelines for surgical techniques are as follows:

The incision and resection should follow the surgical standards of the respective center.

* Careful attention should be given to thorough hemostasis after resection.
* In the intervention group, a vacuum-assisted closure (VAC) system will be used for wound closure.

The VAC system should be applied with a suction pressure of -125mmHg to -75 mmHg. In cases where there is a "Vac on vessel" situation, the suction pressure can be reduced to -25 mmHg.

- The control group will receive primary wound closure via either a single-button suture, continuous su-ture, or staple closure, depending on the center's standard.

Drainages should be placed regularly after primary wound closure.

* For the VAC group, the timing of secondary closure is at the discretion of the surgeon. However, the VAC dressing should not remain in place for more than 7 days.
* Secondary wound closure can be performed using a single-button suture, continuous suture, or stapling. A suction drainage should be placed also after secondary wound closure.

A minimum of 50 patients per study arm will be recruited, resulting in a total of at least 100 participants. All patients undergoing sarcoma surgery at participating sarcoma centers between November 2024 and December 2025 will be screened for inclusion in the study.

1. Inclusion Criteria:

   Patients undergoing resection of soft tissue sarcomas in the lower extremity and groin regions are eligible for inclusion if the following criteria are met:
   * Patients must be over 18 years old.
   * Patients of any gender and background can be included.
   * The largest tumor diameter on imaging must be at least 5 cm. Preoperative imaging is required to assess tumor dimensions.
   * Sarcomas must be located in the lower extremity or groin.
   * Cases must be discussed preoperatively at an interdisciplinary tumor board.
   * Patients must provide informed consent to participate in the study.
2. Exclusion Criteria:

Patients meeting any of the following conditions will be excluded:

* Tumors smaller than 5 cm and superficial masses.
* Patients with local recurrences or prior wound healing complications in the surgical area.
* Patients with ulcerating or infected tumors, or those requiring emergency surgery.
* Other Soft Tissue Tumors such as Kaposi sarcoma.
* for whom direct closure is not possible during the initial surgery due to the extent of resection.

ELIGIBILITY:
Inclusion Criteria:

Patients must be over 18 years old.

* Patients of any gender and background can be included.
* The largest tumor diameter on imaging must be at least 5 cm. Preoperative imaging is required to assess tumor dimensions.
* Sarcomas must be located in the lower extremity or groin.
* Cases must be discussed preoperatively at an interdisciplinary tumor board.
* Patients must provide informed consent to participate in the study.

Exclusion Criteria:

* Tumors smaller than 5 cm and superficial masses.
* Patients with local recurrences or prior wound healing complications in the surgical area.
* Patients with ulcerating or infected tumors, or those requiring emergency surgery.
* Other Soft Tissue Tumors such as Kaposi sarcoma.
* for whom direct closure is not possible during the initial surgery due to the extent of resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound complication | 3 Months
  The primary objective of the study is to compare wound complications after vacuum therapy versus direct closure.
Wound Infection | 3 Months
Wound Seroma | 3 Months
  Seroma in Wound
Lymphatic fistula | 3 Months
  Lymphatic fistula or Drainage secretion of >50ml/24h after 5 postoperative days
Wound Dehiscence | 3 Months
  Wound dehiscence
Revision Surgery or conservative treatment | 3 Months
  If Revision surgery or antibiotic treatment is required due to a wound infection.

SECONDARY OUTCOMES:
Risk factors for wound complications | 3 Months
  In addition, the benefit of using drainage to prevent wound infections will be evaluated. For this, the type of drainage, the location of the drainage, the volume of secretion, and the duration of the drainage will be docu-mented. The impact of different sarcoma entities on the occurrence of wound infections will also be investi-gated.
  The effects of BMI, age, smoking, and pre-existing conditions such as diabetes mellitus, cardiovascular diseases, and immunosuppression will be assessed. A subgroup analysis will be performed to evaluate the relevance of neoadjuvant treatment.
  Furthermore, the influence of factors such as tumor location (differences between groin, thigh, and lower leg) and actual tumor size (differences between 5-10 cm and >10 cm) will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No